CLINICAL TRIAL: NCT04949841
Title: A Phase 3 Extension Trial of DELTA 1 and DELTA 2 to Evaluate the Long-term Safety of a Twice-daily Treatment With Delgocitinib Cream 20 mg/g as Needed for up to 36 Weeks in Adult Subjects With Chronic Hand Eczema (DELTA 3)
Brief Title: Open-label Multi-site Extension Trial in Subjects Who Completed the DELTA 1 or DELTA 2 Trials
Acronym: DELTA 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0133-1403; 2020-002962-15 (EudraCT Number); U1111-1284-2216 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hand Eczema
MeSH Terms: interventions — delgocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- As-needed treatment with delgocitinib (Experimental): Subjects will be treated with delgocitinib cream 20 mg/g twice daily as needed.
  Interventions: Drug: Delgocitinib

INTERVENTIONS:
Drug: Delgocitinib — Delgocitinib cream 20 mg/g

SUMMARY:
The purpose of this extension trial is to evaluate the long-term safety of delgocitinib.

Subjects will visit the clinic every 4 week to assess the safety and efficacy of the treatment, until Week 36. A final follow-up phone call is planned on Week 38.

DETAILED DESCRIPTION:
Subject who completed 16 weeks of treatment with delgocitinib cream 20 mg/g or vehicle cream twice daily in trials DELTA 1 or DELTA 2 will be offered to roll-over to this extension trial.

Subjects will be treated with delgocitinib cream 20 mg/g twice daily only if they need it to control their chronic hand eczema. In the periods when the disease is controlled, no treatment will be administered.

Clinic visits every 4 weeks are planned (with the possibility of unscheduled visits) to investigate safety and efficacy of treatment, as well as its effect on patient-reported outcomes (PROs).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have met eligibility criteria at screening and baseline in the parent trial (DELTA 1 or DELTA 2).
* Participants must have completed the treatment period in the parent trial (to be assessed at baseline visit in this extension trial).
* Participants must have complied with the clinical trial protocol in the parent trial to the satisfaction of the investigator.
* A woman of childbearing potential must use an acceptable method of birth control throughout the trial up until the end-of-treatment/early termination visit.

Exclusion Criteria:

* Participants who prematurely discontinued treatment with IMP or initiated rescue medication in the parent trial.
* Participants who experienced any adverse event (AE) during participation in the parent trial, which precludes further treatment with delgocitinib cream 20 mg/g in the judgement of the investigator.
* Any medical or psychiatric condition that could put the participant at undue risk by participating in the trial, or which, by the investigator's judgment, makes the participant inappropriate for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (85):
- Belgium (6):
  - LEO Investigational Site, Brussels
  - LEO Investigational Site, Ghent
  - LEO Investigational Site, Kortrijk
  - LEO Investigational Site, Leuven
  - LEO Investigational Site, Loverval
  - LEO Investigational Site, Maldegem
- Canada (16):
  - LEO Investigational Site, Calgary, Alberta
  - LEO Investigational Site, Edmonton, Alberta
  - LEO Investigational Site, Surrey, British Columbia
  - LEO Investigational Site, Vancouver, British Columbia
  - LEO Investigational Site, Fredericton, New Bruswick
  - LEO Investigational Site, Ajax, Ontario
  - LEO Investigational Site, Cobourg, Ontario
  - LEO Investigational Site, Etobicoke, Ontario
  - LEO Investigational Site, Hamilton, Ontario
  - LEO Investigational Site, Kingston, Ontario
  - LEO Investigational Site, London, Ontario
  - LEO Investigational Site, Markham, Ontario
  - LEO Investigational Site, Toronto, Ontario
  - LEO Investigational Site, Waterloo, Ontario
  - LEO Investigational Site, Windsor, Ontario
  - LEO Investigational Site, Montreal, Quebec
- Denmark (3):
  - LEO Investigational Site, Aarhus N
  - LEO investigational Site, Copenhagen
  - LEO Pharma Investigational Site, Hellerup
- France (10):
  - LEO Investigational Site, Bordeaux
  - LEO Investigational Site, Dijon
  - LEO Investigational Site, Le Mans
  - LEO Investigational Site, Lille
  - LEO Investigational Site, Martigues
  - LEO Pharma Investigational Site, Nantes
  - LEO Investigational Site, Nice
  - LEO Investigational Site, Paris
  - LEO Investigational Site, Reims
  - LEO Investigational Site, Toulouse
- Germany (20):
  - LEO Investigational Site, Aachen
  - LEO Investigational Site, Bad Bentheim
  - LEO Investigational Site, Berlin
  - LEO Investigational Site, Bretzenheim
  - LEO Investigational Site, Dresden
  - LEO Investigational Site, Frankfurt am Main
  - LEO Investigational Site, Friedrichshafen
  - LEO Investigational Site, Gera
  - LEO Investigational Site, Göttingen
  - LEO Investigational Site, Hamburg
  - LEO Investigational Site, Hanover
  - LEO Investigational Site, Haßfurt
  - LEO Investigational Site, Jena
  - LEO Investigational Site, Lübeck
  - LEO Investigational Site, Mahlow
  - LEO Pharma Investigational Site, Memmingen
  - LEO Investigational Site, München
  - Leo Investigational Site, Münster
  - LEO Investigational Site, Osnabrück
  - LEO Investigational Site, Stuttgart
- Italy (4):
  - LEO Investigational Site, Brescia
  - LEO Investigational Site, L’Aquila
  - LEO Investigational Site, Rome
  - LEO Investigational Site, Vicenza
- Netherlands (5):
  - LEO Investigational Site, Amsterdam
  - LEO Investigational Site, Bergen op Zoom
  - LEO Investigational Site, Groningen
  - LEO Investigational Site, Hoofddorp
  - LEO Investigational Site, Utrecht
- Poland (10):
  - LEO Investigitional Site, Bialystok
  - LEO Investigational Site, Bialystok
  - LEO Investigational Site, Gdansk
  - LEO Investigational Site, Krakow
  - LEO Investigational Site, Lodz
  - LEO Investigational Site, Lublin
  - LEO Investigational Site, Osielsko
  - LEO Pharma Investigational Site, Rzeszów
  - LEO Investigational Site, Warsaw
  - LEO Investigational Site, Wroclaw
- Spain (7):
  - LEO Investigational Site, Alicante
  - LEO Investigational Site, Badalona
  - LEO Investigitional Site, Barcelona
  - LEO Investigational Site, Bilbao
  - LEO Investigational Site, Madrid
  - LEO Investigational Site, Mieres
  - LEO Investigational Site, Seville
- United Kingdom (4):
  - LEO Investigational Sites, Redhill, Surrey
  - LEO Investigational Site, London
  - LEO Investigational Site, Middlesbrough
  - LEO Investigational Site, Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial enrolled subjects who completed one of the 2 pivotal phase 3 trials with delgocitinib cream 20 mg/g or cream vehicle (parent trials - Trial 1401 [NCT04871711] or Trial 1402 [NCT04872101]).
Groups:
- As-needed Treatment With Delgocitinib: Subjects will be treated with delgocitinib cream 20 mg/g twice daily as needed. >
  > Delgocitinib: Delgocitinib cream 20 mg/g
Period: Overall Study
Arm/Group | As-needed Treatment With Delgocitinib
Started | 801
Completed | 664
Not Completed | 137
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 52
Not completed — Pregnancy | 4
Not completed — Lost to Follow-up | 9
Not completed — Lack of Efficacy | 55
Not completed — Various reasons | 9

BASELINE CHARACTERISTICS:
Groups:
- As-needed Treatment With Delgocitinib: Subjects will be treated with delgocitinib cream 20 mg/g twice daily as needed.>
  > Delgocitinib: Delgocitinib cream 20 mg/g
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 735
  >=65 years | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 512
  Male | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 752
  Unknown or Not Reported | 28
Region of Enrollment [Number; unit: participants]
  Canada | 162
  Netherlands | 16
  Belgium | 19
  Denmark | 20
  Poland | 180
  Italy | 40
  United Kingdom | 23
  France | 68
  Germany | 215
  Spain | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events From Baseline up to Week 38
Description: An AE will be considered treatment emergent if it started after the baseline visit
Time Frame: From baseline up to Week 38
Measure: Number; unit: events
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
events | 1238

2. Secondary Outcome: Number of Participants With IGA-CHE Score at Each Scheduled Visit From Baseline up to Week 36
Description: The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: From baseline up to Week 38
Measure: Count of Participants; unit: Participants
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
Participants
  At baseline : 0-Clear | 77
  At baseline : 1- Almost Clear | 83
  At baseline : 2- Mild | 345
  At baseline : 3- Moderate | 243
  At baseline : 4- Severe | 53
  Week 4 : 0-Clear | 58
  Week 4 : 1- Almost Clear | 76
  Week 4 : 2- Mild | 436
  Week 4 : 3- Moderate | 189
  Week 4 : 4- Severe | 28
  Week 8 : 0-Clear | 73
  Week 8 : 1- Almost Clear | 82
  Week 8 : 2- Mild | 413
  Week 8 : 3- Moderate | 167
  Week 8 : 4- Severe | 25
  Week 12 : 0-Clear | 79
  Week 12 : 1- Almost Clear | 76
  Week 12 : 2- Mild | 414
  Week 12 : 3- Moderate | 152
  Week 12 : 4- Severe | 18
  Week 16 : 0-Clear | 79
  Week 16 : 1- Almost Clear | 77
  Week 16 : 2- Mild | 407
  Week 16 : 3- Moderate | 147
  Week 16 : 4- Severe | 13
  Week 20 : 0-Clear | 72
  Week 20 : 1- Almost Clear | 90
  Week 20 : 2- Mild | 401
  Week 20 : 3- Moderate | 123
  Week 20 : 4- Severe | 19
  Week 24 : 0-Clear | 65
  Week 24 : 1- Almost Clear | 67
  Week 24 : 2- Mild | 415
  Week 24 : 3- Moderate | 118
  Week 24 : 4- Severe | 15
  Week 28 : 0-Clear | 68
  Week 28 : 1- Almost Clear | 79
  Week 28 : 2- Mild | 408
  Week 28 : 3- Moderate | 109
  Week 28 : 4- Severe | 8
  Week 32 : 0-Clear | 71
  Week 32 : 1- Almost Clear | 67
  Week 32 : 2- Mild | 395
  Week 32 : 3- Moderate | 118
  Week 32 : 4- Severe | 12
  Week 36 : 0-Clear | 115
  Week 36 : 1- Almost Clear | 124
  Week 36 : 2- Mild | 300
  Week 36 : 3- Moderate | 111
  Week 36 : 4- Severe | 13

3. Secondary Outcome: Number of Participants With IGA-CHE Score of 0 (Clear) or 1 (Almost Clear) at Each Scheduled Visit From Baseline up to Week 36.
Description: as for outcome 2
Time Frame: From baseline up to Week 38
Measure: Count of Participants; unit: Participants
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
Participants
  Baseline | 160
  Week 4 | 134
  Week 8 | 155
  Week 12 | 155
  Week 16 | 156
  Week 20 | 162
  Week 24 | 132
  Week 28 | 147
  Week 32 | 138
  Week 36 | 239

4. Secondary Outcome: HECSI Score at Each Scheduled Visit From Baseline up to Week 36
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score).
Time Frame: From baseline up to Week 38
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
score on a scale
  Baseline | 30.8 (36.5)
  Week 4 | 24.3 (27.2)
  Week 8 | 21.4 (25.3)
  Week 12 | 20.2 (23.9)
  Week 16 | 17.9 (21.1)
  Week 20 | 17.8 (22.5)
  Week 24 | 17.7 (19.6)
  Week 28 | 16.6 (19.0)
  Week 32 | 16.9 (20.0)
  Week 36 | 15.4 (20.6)

5. Secondary Outcome: Number of Participants With HECSI-75 at Each Scheduled Visit From Baseline up to Week 36
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score). HECSI-75 is defined as at least 75% improvement in HECSI score from parent trial baseline.
Time Frame: From baseline up to Week 38
Measure: Count of Participants; unit: Participants
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
Participants
  At baseline | 347
  Week 4 | 391
  Week 8 | 415
  Week 12 | 411
  Week 16 | 432
  Week 20 | 438
  Week 24 | 409
  Week 28 | 414
  Week 32 | 411
  Week 36 | 452

6. Secondary Outcome: Number of Participants With HECSI-90 at Each Scheduled Visit From Baseline up to Week 36
Description: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales. The HECSI score will range from 0 (lowest possible score) to 360 (highest possible score). HECSI-90 is defined as at least 90% improvement in HECSI score from parent trial baseline.
Time Frame: From baseline up to Week 38
Measure: Count of Participants; unit: Participants
Arm/Group | As-needed Treatment With Delgocitinib
Number analyzed (Participants) | 801
Participants
  At baseline | 207
  Week 4 | 195
  Week 8 | 224
  Week 12 | 222
  Week 16 | 229
  Week 20 | 239
  Week 24 | 204
  Week 28 | 236
  Week 32 | 220
  Week 36 | 291

ADVERSE EVENTS:
Time Frame: From baseline to week 36
Groups:
- As-needed Treatment With Delgocitinib: As-needed treatment with Delgocitinib cream 20 mg/g (N=801)
Arm/Group | As-needed Treatment With Delgocitinib
All-Cause Mortality (participants affected / at risk) | 3/801
Serious Adverse Events (participants affected / at risk) | 27/801
Other Adverse Events (participants affected / at risk) | 329/801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As-needed Treatment With Delgocitinib (N=801)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Paranasal sinus abscess (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sinusitis aspergillus (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As-needed Treatment With Delgocitinib (N=801)
COVID-19 (Infections and infestations) | 134 (138)
Influenza (Infections and infestations) | 28 (28)
Nasopharyngitis (Infections and infestations) | 128 (161)
Upper respiratory tract infection (Infections and infestations) | 32 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20)
Headache (Nervous system disorders) | 22 (27)
Eczema (Skin and subcutaneous tissue disorders) | 17 (21)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 30 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor seeks publication of all clinical trials in peer-reviewed journals within 12 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by the sponsor within these 12 months, the investigator has the right to publish the results from clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04949841/Prot_SAP_000.pdf